CLINICAL TRIAL: NCT04152928
Title: Applying PET/MR in Neuroendocrine Tumors - Imaging Dynamic Processes in Both Modalities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-19-ES-0582-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuroendocrine Tumors Patients (Experimental): Patients with confirmed NET
  Interventions: Diagnostic Test: PET/MR scan

INTERVENTIONS:
Diagnostic Test: PET/MR scan — The patient will be positioned in the PET/MR with the field of view of the PET including the abdomen, and IV administration of 68Ga-DOTATATE will take place, with initiation of dynamic PET simultaneous with start of IV injection. Dynamic PET imaging will consist of 22 time frames of increasing durations (6 x 10, 3 x 20, 3 x 60, 5 x 180, and 5 x 300 s). The dynamic PET examination will be followed by a whole-body PET/MR scan ranging from the proximal femur to the base of the skull (3 min per bed position) starting at 60 min after injection. MR will be used for attenuation correction of the PET images of the abdomen/pelvis and whole-body. MR protocol will include three plane fast spin echo T2 weighted, DWI, DCE and ASL. The addition of PET/MR to the standard use of PET/CT adds no radiation exposure.

SUMMARY:
Neuroendocrine tumors (NET's) are characterized, among other features, by presence of high concentration of somatostatin receptors. In recent years, for purposes of Positron Emission Tomography (PET) imaging, somatostatin receptor ligands have been labelled with the positron emitting radioisotope 68Ga to form molecules that bind to these somatostatin receptors that are present in high concentration in NET's and in low concentrations, if at all, in normal tissues. In the last 10-15 years, radioactively labelled versions of these molecules have been used for both diagnostic and therapeutic purposes in the management of patients with NET's.

The main goal of this study is to assess the feasibility of performing dynamic 68Ga-DOTATATE PET in the PET/MRI system and analyzing the effect of diffusion and perfusion over Ki values.

DETAILED DESCRIPTION:
Working hypotheses

1. The PET/MR system will provide dynamic PET images of at least comparable quality compared to PET/CT. Dynamic PET/MR will be feasible, with the 45 minute dynamic PET acquisition occurring during the MR sequences, eliminating the need for the patient to undergo two separate lengthy studies.
2. Diffusion and perfusion parameters extracted from MRI sequences will provide information that improves the process of Ki evaluation.
3. The use of advanced statistics methodologies, such as those used in radiomics, to correlate Ki data with diffusion and perfusion data will provide a quantification tool that will improve staging, prediction and monitoring after treatment.
4. Parametric Patlak Ki images calculated from the dynamic series of PET images will show better contrast between tumors and normal tissue, as compared to contrast in the conventional static images obtained from the last time frame of the dynamic image series. Tumors identified on the static PET image will be visualized at least as well on Patlak Ki images, and possibly additional tumor foci may be identified. MRI should assist in confirming and interpreting such findings.

Research plan Population: 50 patients with NETs that have evidence of at least one abdominal lesion with diameter greater than 2cm. All patients will be aged 18 years or older of both sexes.

Inclusion criteria: Patients with confirmed NET. Exclusion criteria: Patients younger than 18 years; pregnancy; other known active malignancy; contraindication to MRI tests or intravenous contrast agents.

ELIGIBILITY:
Inclusion Criteria:

1.Patients with confirmed NET.

Exclusion Criteria:

1. Patients younger than 18 years.
2. Patients pregnancy.
3. Patients with other known active malignancy.
4. Patients contraindication to MRI tests or intravenous contrast agents.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-25 (Estimated); Primary Completion 2021-03-25 (Estimated); Study Completion 2022-02-25 (Estimated)

PRIMARY OUTCOMES:
Patients who performing dynamic 68Ga-DOTATATE PET in the PET/MRI system and analyzing the effect of diffusion and perfusion over Ki values. | 1 year

IPD SHARING:
Plan to Share IPD: Undecided